CLINICAL TRIAL: NCT01892488
Title: Randomized Double Blind Placebo-controlled Study to Demonstrate That Antibiotics Are Not Needed in Moderate Acute Exacerbations of COPD - The ABACOPD Study
Brief Title: Study to Demonstrate That Antibiotics Are Not Needed in Moderate Acute Exacerbations of COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: CAPNETZ Stiftung (Other)
Responsible Party: Principal Investigator, Tobias Welte, Prof. Dr., Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol-Code: 002/2012; 2012-003234-16 (EudraCT Number)
Record Dates: First submitted 2013-06-27; First posted 2013-07-04 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; AE-COPD; Chronic obstructive pulmonary disease; acute exacerbations of Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — sultamicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lactose pill (Placebo Comparator): Placebo for 5 days as supplement to standard of care for patients with AE-COPD
  Interventions: Drug: Placebo
- Sultamicillin (Experimental): Antibiotic therapy with aminopenicillin + betalactamase inhibitor (oral Sultamicillin (2 x 750mg)) for 5 days as supplement to standard of care for patients with AE-COPD
  Interventions: Drug: Sultamicillin

INTERVENTIONS:
Drug: Sultamicillin — Standard of care: Each patient will receive inhaled fast-acting bronchodilators (up to a maximum of 4 - 6 times daily 2 puffs (100µg) of salbutamol or other equivalent inhaled fast-acting bronchodilators), systemic corticosteroids (prednisolone 40mg/d p.o. for 7 - 10 days) and oxygen in case of hypoxemia in a standardized fashion. The pre-existing COPD medication will be continued as indicated.
  Experimental intervention:
  Antibiotic therapy with aminopenicillin + betalactamase inhibitor (oral Sultamicillin (2 x 750mg)) for 5 days as supplement to standard of care for patients with AE-COPD.
  Other Names: aminopenicillin + betalactamase inhibitor
  Arms: Sultamicillin
Drug: Placebo — Standard of care: Each patient will receive inhaled fast-acting bronchodilators (up to a maximum of 4 - 6 times daily 2 puffs (100µg) of salbutamol or other equivalent inhaled fast-acting bronchodilators), systemic corticosteroids (prednisolone 40mg/d p.o. for 7 - 10 days) and oxygen in case of hypoxemia in a standardized fashion. The pre-existing COPD medication will be continued as indicated.
  Control intervention:
  Placebo for 5 days as supplement to standard of care for patients with AE-COPD
  Other Names: Placebo: Lactose pill
  Arms: lactose pill

SUMMARY:
The ultimate goal is to reduce unnecessary antibiotic prescriptions which drive the development of antibiotic resistance in the community. The primary objective of ABACOPD is to demonstrate in a sufficiently sized clinical study that there is no relevant increase in the "failure-rate" for patients with acute moderate exacerbations of COPD (AE-COPD) treated with placebo instead of antibiotic treatment both on top of standard of care. A patient is classified as treatment failure if additional antibiotic therapy is required during treatment period or until the test of cure visit (TOC at day 30, primary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Adults, either sex, older or equal than 40 years of age
* For female patients, the following conditions are to be met:

  * has been postmenopausal for at least 1 year, or
  * is surgically incapable of bearing children, or
  * is of childbearing potential, and the following conditions are met:

    * has a negative pregnancy test (urine- or serum-based) immediately before study entry (i.e., before the start of treatment or any other study procedure that could potentially harm the fetus), and one or more of following criteria
    * must agree to abstinence or use an accepted method of contraception. The subject must agree to continue with the same method throughout the study.
    * having only female sexual partners
    * sexual relationship with sterile male partners only
* Patients diagnosed with COPD stages I-IV as defined by the Global initiative for chronic Obstructive Lung disease (GOLD).

and

* Doctor's diagnosis of acute (onset < 7 days) moderate exacerbation of COPD defined by a sustained worsening of the patient's condition (including at least 2 of the following symptoms: increased dyspnea, increased sputum production, sputum purulence and increased cough), from the stable state and beyond normal day-to-day variations, necessitating a change in regular medication in patient with underlying COPD, needing additional medical assistance.
* Absence of community acquired pneumonia or lower respiratory tract infection with a clear indication for antibiotic treatment as determined by Procalcitonin level < 0.25 ng/mL and/or absence of pulmonary infiltrates on routine chest x-ray.
* Smoking history of at least 10 Pack Years or more.
* Patients must be able to complete diaries and quality of life questionnaires.
* Patients must sign and date an informed consent prior to any study procedures.

Exclusion Criteria:

* Severe exacerbation: defined by need for ventilatory support (indicated by severe dyspnea with failure to respond to emergency treatment and/or persistent hypoxemia (PaO2 <50 mm Hg despite O2 administration and / or respiratory acidosis (pH <7.35 and PaCO2> 45mmHg)) or mental confusion or circulatory insufficiency (need of vasopressors)
* Fever (>38.5°C)
* Known impaired hepatic or renal function
* Active or suspected tuberculosis infection of the respiratory tract
* Acute exacerbation of asthma
* Suspected or known hypersensitivity to, or suspected serious adverse reaction to sultamicillin; suspected or known hypersensitivity to penicillins or cephalosporins
* Immunosuppression or Immunosuppressive therapy (cytostatic chemotherapy within last 28 days or neutropenia (neutrophils < 1000/µ)l; systemic corticosteroids (≥20 mg prednisolon equivalent/day > 14 days; HIV-infection; immunosuppression after organ- or bone marrow transplant)- Patients with metastatic or hematological malignancy, splenectomized patients or patients with known hyposplenia or asplenia
* Oral/parenteral antibiotic use within 30 days prior to randomization (a singular administration of antibiotics prior to randomization is allowed)
* In-patient treatment within the last 30 days
* An antibiotic is clearly indicated for treatment of a known infection
* Known MRSA (methicillin-resistant Staphylococcus aureus) colonization or infection
* Patients with known bronchiectasis
* Patients with known bacterial airway colonization (>3 positive sputum cultures in the previous year)
* Progressively fatal disease, or life expectancy ≤6 months
* Mononucleosis
* Lymphatic leukemia
* Severe gastro-intestinal disorders with vomiting and diarrhea
* Women who are breast feeding
* Patients who have received treatment with any other investigational drug within 1 month prior to study entry, or have such treatment planned for the study period during treatment and follow up phase.
* Patients with mental conditions rendering them unable to understand the nature, scope, and possible consequences of the study.
* Patients unlikely to comply with the protocol, e.g., uncooperative attitude, inability to return for follow up visits, and unlikelihood of completing the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2013-06-07 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Additional antibiotic therapy to study medication during treatment period or until the test of cure visit (at day 30) | up to day 30
  Assessment of additional antibiotic therapy:
  Patients will be asked at every visit about use of additional antibiotic therapy. In the case of use of additional antibiotic therapy the exact starting date, the active compound, the dose administered, the route of administration,the length of treatment and the indication will be registered. Only additional antibiotic therapy for AE-COPD will be counted as treatment failure.

SECONDARY OUTCOMES:
To evaluate long-term consequences of Placebo treatment | up to 1 year
  * Relapse rate
  * Time to relapse
To assess patient's clinical improvement relative to treatment | up to 30 days
  * Clinical cure rate at the "end of therapy visit" (at day 6)
  * Clinical cure rate at the "test Of cure visit" (at day 30) (both determined by patient-centered outcomes (diary cards))
To assess additional efficacy endpoints and health outcome evaluations | up to 1 year
  * Changes in COPD Assessment Test(CAT)
  * Changes in Exacerbations of Chronic Pulmonary Disease Tool-Patient reported outcome (EXACT-PRO)
  * Additional antibiotic therapy
  * Time to next exacerbation
  * Number of exacerbations during follow up
  * Per-subject relapse rate at the LFU (Late Follow Up) visits in the subset of subjects in the CE population who were clinically cured at the TOC visit
  * Changes in length of stay in hospital for hospitalized patients
  * All cause mortality

OTHER OUTCOMES:
Assessment of safety: | up to 1 year
  Key criteria for safety are:
  adverse events, serious adverse events, changes in physical examination, vital signs, laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Gernot Rohde, Prof. Dr., Study Director — CAPNETZ Stiftung; Tobias Welte, Prof.Dr., Principal Investigator — Hannover Medical School
Locations (32):
- Germany (32):
  - Universitätsklinikum Aachen, Aachen
  - Krankenhaus Bad Arolsen, Bad Arolsen
  - Lungenklinik Ballenstedt, Ballenstedt
  - Charité - Universitätsmedizin Berlin, Berlin
  - HELIOS Klinikum Emil von Behring Berlin, Berlin
  - Pneumologische Praxis am Schloss Charlottenburg Berlin, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Klinikum der Ruhr-Universität Bochum, Bochum
  - Pneumologische Gemeinschaftspraxis Bonn, Bonn
  - Forschungszentrum Borstel, Borstel
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitätsklinikum Dresden, Dresden
  - Pneumologische Klinik Waldhof Elgershausen, Elgershausen
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Praxis Dr. med. Ina Itzigehl Euskirchen, Euskirchen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Greifswald, Greifswald
  - HELIOS Klinik Hagen-Ambrock, Hagen
  - Elbpneumologie Hamburg, Hamburg
  - Schwerpunktpraxis Colonnaden Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhausen
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein Kiel, Kiel
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Diakoniekrankenhaus Rotenburg, Rotenburg (Wümme)
  - Krankenhaus Bethanien Solingen, Solingen
  - HELIOS Klinikum Wuppertal-Barmen, Wuppertal

REFERENCES:
- [Derived] Rohde GG, Koch A, Welte T; ABACOPD study group. Randomized double blind placebo-controlled study to demonstrate that antibiotics are not needed in moderate acute exacerbations of COPD--the ABACOPD study. BMC Pulm Med. 2015 Jan 27;15:5. doi: 10.1186/1471-2466-15-5. PMID 25623589